CLINICAL TRIAL: NCT04988360
Title: VRx@Home: Pilot RCT to Evaluate the Effectiveness of Immersive Virtual Reality Therapy on People With Dementia Living at Home
Brief Title: VRx@Home: Study to Evaluate VR-therapy for PwD Living at Home
Acronym: VRx@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other)
Responsible Party: Principal Investigator, Lora Appel, Post-doc Research Fellow; Assistant Professor, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: VRx@Home Pilot
Record Dates: First submitted 2021-06-21; First posted 2021-08-03 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Dementia
Keywords: Virtual Reality; Tablets; Interpersonal Relations; Community Health Services; Apathy; Depressive Symptoms; Behavioral Symptoms; Quality of Life; Caregivers; Spouse Caregivers; Family Caregivers
MeSH Terms: conditions — Dementia; Lethargy; Depression; Behavioral Symptoms | interventions — Smart Glasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: HMD first (Experimental): Those assigned to group A will use the head-mounted display (HMD) VR intervention first. Caregivers will be trained to use the HMD-system and asked to use that system for the duration of T1 (weeks 1 & 2). At the end of T1 they will be asked to complete standardized questionnaires and will participate in a semi-structured interview about their experiences. At the beginning of T2 (weeks 3 & 4), they will then be trained to use the tablet-system, which will be used for the duration of T2. At the completion of T2, the dyad will again complete the same standardized questionnaires and will participate in a semi-structured interview about their experiences. Each session is expected to include 20 minutes of VR exposure. Each session throughout T1 and T2 is to be video-recorded by the caregiver-participant so that reactions and interactions can later be analyzed.
  Interventions: Device: HMD: Immersive VR; Device: Tablet: Non-immersive VR
- Group B: Tablet first (Experimental): Those assigned to group B will use the tablet VR intervention first. Caregivers will be trained to use the tablet-system and asked to use that system for the duration of T1 (weeks 1 & 2). At the end of T1 they will be asked to complete standardized questionnaires and will participate in a semi-structured interview about their experiences. At the beginning of T2 (weeks 3 & 4), they will then be trained to use the HMD-system, which will be used for the duration of T2. At the completion of T2, the dyad will again complete the same standardized questionnaires and will participate in a semi-structured interview about their experiences. Each session is expected to include 20 minutes of VR exposure. Each session throughout T1 and T2 is to be video-recorded by the caregiver-participant so that reactions and interactions can later be analyzed.
  Interventions: Device: HMD: Immersive VR; Device: Tablet: Non-immersive VR

INTERVENTIONS:
Device: HMD: Immersive VR — Participants with dementia will view 360-degree films using a commercially-available Virtual Reality head mounted display (HMD) that has built-in speakers. While wearing the HMD, participants with dementia will be able to visually explore the virtual environments by turning their head to face different directions. Caregivers-participants will take part in the VR experience concurrently by viewing a tablet that is connected to the HMD through the "screen mirroring" function.
  Other Names: Head-mounted display; Headset
Device: Tablet: Non-immersive VR — Participants with dementia will view 360-degree films on a commercially-available tablet that has built-in speakers. Participants with dementia will be able to visually explore the virtual environment using the touch screen (dragging the view around with one's finger). Caregiver-participants will take part in the VR experience concurrently by viewing the tablet while sitting or standing beside the participant with dementia.

SUMMARY:
The investigators are designing and rigorously evaluating the first Virtual Reality-therapy program for people with dementia (PwD) living at home, administered by their informal caregivers (family/friends). Virtual Reality (VR) presents a unique opportunity to transport people to a world outside of their confined spaces, into calming and stimulating settings (lush forest, peaceful beach, cheerful playground). Virtual Reality-therapy is a non-pharmacological approach that uses VR "experiences'' to stimulate brain function, improve psychological health, engage, and relax. It has potential to reduce symptoms of dementia such as apathy, depression, loneliness, sundowning, and the use of sedating medications with known negative side-effects.

Caregivers of PwD are more likely to feel worried, tired, overwhelmed, and depressed than non-PwD caregivers. Symptoms of dementia and caregiver stress often result in early institutionalization of PwD; management of challenging symptoms may help PwD remain in their homes for longer while improving their, and their caregivers', Quality of Life (QoL). Addressing the wellbeing of caregivers is an often overlooked, yet integral part of interventions for PwD. It ensures intervention feasibility but also has a distinct impact on our system, reducing healthcare needs of caregivers and allowing them to continue contributing as caregivers.

In this pilot study the investigators will train and assist caregivers to conduct Virtual Reality-therapy with their loved-ones at home using two devices: a head-mounted display and a tablet. This pilot study will assess: (1) the acceptability of the VR devices (2) feasibility of the study methods, (3) the impact of VR-therapy on PwD and caregiver outcomes. These findings will be used to inform a future randomized controlled trial (RCT).

DETAILED DESCRIPTION:
This pilot trial will be a mixed-methods, parallel arm RCT with a target total recruitment of 30 participants (15 dyads of PwD and caregivers). Each dyad will participate in the study for a total of 4 weeks.

After obtaining informed consent, the research coordinator will set up a time convenient to both parties (the researcher and participant dyad) to conduct a baseline semi-structured interview that collects demographics as well as a questionnaire consisting of validated instruments on the outcome measures of interest (e.g. quality of life, apathy, etc.) Once baselines data collection is complete, the dyad will be randomized into one of two study arms, determining which VR technology they will be using first: (A) HMD first (immersive VR), or (B) Tablet first (non-immersive VR). Those assigned to Group A will use the HMD for weeks 1-2 and the tablet for weeks 3-4. Those assigned to Group B will use the tablet for weeks 1-2 and the HMD for weeks 3-4. After randomization, the participants, caregivers, and research personnel will not be blind to treatment allocation given the nature of the interventions.

The benefits of this randomized crossover design include the: (1) ability to compare the outcomes between immersive VR (HMD system) and non-immersive VR (tablet-only system) where each dyad serves as their own control, reducing the effects of inter-individual variability or disease progression, (2) opportunity for all participants to use the VR HMD, and (3) ability to explore whether the intervention "washes-out" soon after each therapy period or if it has a carryover effect.

Irrespective of experimental arm (Group A or Group B), the intervention consists of therapy sessions administered five times per week, at times agreeable to the dyad, for a total of approximately 80 minutes per week (20 minutes per viewing, 4 times per week). Prior to each session, the caregiver-participant will commence video-recording via the video-conferencing application (as taught during the training session). Once the recording is confirmed, the participants may start their session. During each session, PwD should be seated in a comfortable and secure chair of their choice. Caregiver-participants will help PwD equip the device and launch the films. The participant dyad will be able to select from a wide range of films available on each device. Once the selected film starts to play, the caregiver-participant will be seated nearby to ensure the safety of the PwD and to jointly experience VR. Once the dyad has finished using VR and their discussions/interactions about VR have concluded, the caregiver-participant may stop the video recording. The video recording will be stored securely automatically. Each member of the study dyad will then complete a personal reflection about the study session.

In addition to the video-recording (used to analyze participant interaction and conduct conversation analysis) some data collection tools are meant to be filled in after each session. The remaining data is collected via a structured questionnaire containing validated instruments and open-ended questions filled in at Baseline (T0), at the end of Weeks 1-2 (T1), and at the end of Weeks 3-4 (T2), to gather experiences using both the VR and tablet devices, and potential impact on clinical outcomes. The usability of each VR technology will be assessed at the end of T1 and T2.

ELIGIBILITY:
PwD inclusion criteria:

* Individuals who are 65 years of age or older.
* Individuals living at home with a family caregiver.
* Individuals diagnosed with mild to moderate dementia.

PwD exclusion criteria:

* Individuals with open wounds on face (sutured lacerations exempted).
* Individuals with a history of seizures or epilepsy.
* Individuals with a pacemaker.
* Individuals with head trauma or stroke leading to their current admission.
* Individuals with cervical conditions or injuries that would make it unsafe for them to use the VR headset.
* Individuals with alcohol related dementia/ Korsakoff syndrome.
* Individuals who have a Public Guardian and Trustee (PGT) as Substitute Decision Maker (SDM).
* Individuals who cannot speak and understand English

Caregiver inclusion criteria:

* Live with a PwD
* Identify as a primary caregiver for the PwD

Caregiver exclusion criteria:

* Individuals who cannot speak and understand English
* Individuals who are professional/formal caregivers for the PwD
* Individuals who are cognitively unable to provide informed consent for themselves

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Usability scores of first VR intervention used | Day 14 of participation
  System Usability Scale (SUS) will be administered to evaluate device usability/ease-of-use of the first type of VR intervention used during the study: head-mounted device (HMD) for participant group A, and tablet for participant group B). Each participant (caregiver and person with dementia) will complete this questionnaire after 2 weeks of using the respective VR intervention. The SUS is a 10-item questionnaire employing 5-point Likert scales. Calculated scores range from 0-100. Higher scores indicate better system usability.
Usability scores of second VR intervention used | Day 28 of participation
  System Usability Scale (SUS) will be administered to evaluate device usability/ease-of-use of the second type of VR intervention used during the study: head-mounted device (HMD) for participant group B, and tablet for participant group A. Each participant (caregiver and person with dementia) will complete this questionnaire after 2 weeks of using the respective VR intervention. The SUS is a 10-item questionnaire employing 5-point Likert scales. Calculated scores range from 0-100. Higher scores indicate better system usability.
Appropriateness of the study procedures for feasible use of VR-therapy in the home using first intervention | Day 14 of participation
  Semi-structured interview questions will assess opinions on the devices and VR-therapy program experience including: (1) Device comfort, (2) Device tolerance, (3) Content preferences, (4) Challenges, (5) Areas for program improvement, (6) Willingness to continue to use VR, (7) Willingness to recommend VR to others, (8) Open-ended question to capture any other opinions or concerns. Both participants (caregiver and person with dementia) will also complete informal personal reflections about the sessions to capture any feelings, observations, or opinions about VR or the study procedures not otherwise collected by the study tools.
Appropriateness of the study procedures for feasible use of VR-therapy in the home using second intervention | Day 28 of participation
  Semi-structured interview questions will assess opinions on the devices and VR-therapy program experience including: (1) Device comfort, (2) Device tolerance, (3) Content preferences, (4) Challenges, (5) Areas for program improvement, (6) Willingness to continue to use VR, (7) Willingness to recommend VR to others, (8) Open-ended question to capture any other opinions or concerns. Both participants (caregiver and person with dementia) will also complete informal personal reflections about the sessions to capture any feelings, observations, or opinions about VR or the study procedures not otherwise collected by the study tools.

SECONDARY OUTCOMES:
Change from baseline perceived relationship quality within the participant dyad scores | Days 1, 14, and 28 of participation
  The Dyadic Relationship Scale (DRS) will be completed by both participants (caregiver and person with dementia) to evaluate the perceived quality of the dyad relationship. The DRS is an 11-item questionnaire employing 4-point Likert scales. The DRS contains two subscales: Positive Dyadic Interaction and Dyadic Strain. Scores for the Positive Dyadic Interaction subscale range from 6-24, where higher scores indicate more positive dyadic interaction. Scores for the Dyadic Strain subscale range from 5-20, where higher scores indicate higher levels of dyadic strain.
Change from baseline apathy scores in participants with dementia | Days 1, 14, and 28 of participation
  The Apathy Evaluation Scale (AES) and will be completed by both participants (caregiver and person with dementia) to determine convergence/divergence of scores. The AES is an 18-item questionnaire employing 4-point Likert scales. Scores range from 18-72. Higher scores indicate more apathy.
Change from baseline depression scores in participants with dementia | Days 1, 14, and 28 of participation
  The Depression Cornell Scale for Depression in Dementia (CSDD) and will be completed by caregiver-participants. The CSDD is a 19-item questionnaire employing 3-point Likert scales and an "unable to evaluate" option. Scores range from 0-38. Higher scores indicate greater signs of depression.
Change from baseline depression scores in participants with dementia | Days 1, 14, and 28 of participation
  The Short Geriatric Depression Scale (GDS) and will be completed by participants with dementia. The GDS is a 15-item questionnaire employing "yes/no" options that may be used with older adults with mild to moderate cognitive impairment. Scores range from 0-15. Higher scores indicate greater signs of depression.
Change from baseline behavioural disturbance scores in participants with dementia | Days 1, 14, and 28 of participation
  Behavioural symptoms related to cognition, functional autonomy, somatic symptoms, and psychiatric symptoms displayed by participants with dementia will be evaluated by the Dementia Behaviour Disturbance Scale (DBD) which will be completed by caregiver-participants. The DBD is a 28-item questionnaire employing 5-point Likert scales. Scores range from 0-112. Higher scores indicate greater behavioural disturbance.
Change from baseline quality of life (QoL) scores for participants with dementia as assessed by the BASQID. | Days 1, 14, and 28 of participation
  The Bath Assessment of Subjective Quality of Life in Dementia (BASQID) will be administered to evaluate the subjective quality of life of participants with dementia. The BASQID is a 14-item questionnaire employing 5-point Likert scales and contains two subscales Life Satisfaction (LS) and Feelings of Positive Quality of Life (FPQ) . Calculated scores range from 0-100. Higher scores indicate greater subjective quality of life.
Change from baseline quality of life (QoL) scores for participants with dementia and caregiver-participants as assessed by the QoL-AD | Days 1, 14, and 28 of participation
  The Quality of Life in Alzheimer's Dementia (QoL-AD) will be administered to participants with dementia and caregiver-participants to evaluate subjective quality of life. The QoL-AD is a 13-item questionnaire employing 4-point Likert scales. Calculated scores range from 0-52. Higher scores indicate greater subjective quality of life.
Change from baseline wellbeing scores for participants with dementia and caregiver-participants as assessed by the WHO (Five) Well-Being Index | Days 1, 14, and 28 of participation
  The WHO (Five) Well-Being Index will be administered to participants with dementia and caregiver-participants to evaluate subjective wellbeing. The WHO (Five) is a 5-item questionnaire employing 6-point Likert scales. Calculated scores range from 0-25. A score of 0 represents the worst possible and a score of 25 represents the best possible quality of life. A score below 13 represents poor wellbeing. A change of 10% represents a significant change in wellbeing.
Change from baseline quality of life (QoL) scores for caregiver-participants as assessed by the Caregiver Self-Assessment Questionnaire | Days 1, 14, and 28 of participation
  The Caregiver Self-Assessment Questionnaire will be completed by caregiver-participants and will be used to evaluate the subjective quality of life (QoL) of caregiver-participants. This scale contains 16 "Yes/No" questions and 2 visual analog scales (VAS) ranging from 1-10. Total scores range from 2-36. Higher scores indicate lower subjective caregiver quality of life.
Change from baseline quality of life (QoL) scores for caregiver-participants as assessed by the CarerQoL-7D and CarerQoL-VAS | Days 1, 14, and 28 of participation
  The CarerQoL-7D (CarerQol instrument which measures the impact of informal care on seven important burden dimensions and values this in terms of general quality of life, and the CarerQoL-VAS (Visual Analog Scale) will be completed by caregiver-participants and will be used to evaluate the subjective quality of life (QoL) of caregiver-participants. The CarerQoL-7D is a 7-item questionnaire employing 3-point Likert scales that provides a comprehensive description of the caregiving situation. The CarerQoL-VAS is a VAS ranging from 0-10 that provides a valuation of informal care in terms of well-being. The CarerQoL-VAS is an optional addition to the CarerQoL-7D and is not used when calculating scores. Calculated QoL scores range from 0-100 where higher scores indicate better caregiving situations.
Change from baseline feelings of caregiver reward for caregiver-participants | Days 1, 14, and 28 of participation
  The Positive Aspects of Caregiving (PAC) tool will be completed by caregiver-participants and will be used to evaluate subjective positive feelings associated with being a caregiver for the person with dementia. The PAC is a 9-item questionnaire that measures feelings of reward in Alzheimer's caregiving and has two subcomponents: self affirmation and outlook on life. Total scores range from 9-45 where higher scores indicate greater feelings of caregiver reward.
Change from baseline feelings of caregiver burden for caregiver-participants | Days 1, 14, and 28 of participation
  The Short Zarit Burden Interview tool will be completed by caregiver-participants and will be used to evaluate subjective feelings of caregiver burden associated with being a caregiver for the person with dementia. The Short Zarit Burden Interview is a 6-item questionnaire that employs a 5-point Likert scale. Total scores range from 0-24 where higher scores indicate greater feelings of caregiver burden.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Acclaim Health, Oakville, Ontario
  - Circle of Care, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appel L, Appel E, Bogler O, Wiseman M, Cohen L, Ein N, Abrams HB, Campos JL. Older Adults With Cognitive and/or Physical Impairments Can Benefit From Immersive Virtual Reality Experiences: A Feasibility Study. Front Med (Lausanne). 2020 Jan 15;6:329. doi: 10.3389/fmed.2019.00329. eCollection 2019. PMID 32010701
- [Background] Appel L, Kisonas E, Appel E, Klein J, Bartlett D, Rosenberg J, Smith C. Introducing virtual reality therapy for inpatients with dementia admitted to an acute care hospital: learnings from a pilot to pave the way to a randomized controlled trial. Pilot Feasibility Stud. 2020 Oct 31;6(1):166. doi: 10.1186/s40814-020-00708-9. PMID 33292729
- [Background] Appel L, Kisonas E, Appel E, Klein J, Bartlett D, Rosenberg J, Smith CN. Administering Virtual Reality Therapy to Manage Behavioral and Psychological Symptoms in Patients With Dementia Admitted to an Acute Care Hospital: Results of a Pilot Study. JMIR Form Res. 2021 Feb 3;5(2):e22406. doi: 10.2196/22406. PMID 33533720
- [Background] Berman MG, Kross E, Krpan KM, Askren MK, Burson A, Deldin PJ, Kaplan S, Sherdell L, Gotlib IH, Jonides J. Interacting with nature improves cognition and affect for individuals with depression. J Affect Disord. 2012 Nov;140(3):300-5. doi: 10.1016/j.jad.2012.03.012. Epub 2012 Mar 31. PMID 22464936
- [Background] Brodaty H, Donkin M. Family caregivers of people with dementia. Dialogues Clin Neurosci. 2009;11(2):217-28. doi: 10.31887/DCNS.2009.11.2/hbrodaty. PMID 19585957
- [Background] Diette GB, Lechtzin N, Haponik E, Devrotes A, Rubin HR. Distraction therapy with nature sights and sounds reduces pain during flexible bronchoscopy: a complementary approach to routine analgesia. Chest. 2003 Mar;123(3):941-8. doi: 10.1378/chest.123.3.941. PMID 12628899
- [Background] Hughes JC, Louw SJ. Electronic tagging of people with dementia who wander. BMJ. 2002 Oct 19;325(7369):847-8. doi: 10.1136/bmj.325.7369.847. No abstract available. PMID 12386013
- [Background] Morita E, Fukuda S, Nagano J, Hamajima N, Yamamoto H, Iwai Y, Nakashima T, Ohira H, Shirakawa T. Psychological effects of forest environments on healthy adults: Shinrin-yoku (forest-air bathing, walking) as a possible method of stress reduction. Public Health. 2007 Jan;121(1):54-63. doi: 10.1016/j.puhe.2006.05.024. Epub 2006 Oct 20. PMID 17055544
- [Background] Park BJ, Tsunetsugu Y, Kasetani T, Kagawa T, Miyazaki Y. The physiological effects of Shinrin-yoku (taking in the forest atmosphere or forest bathing): evidence from field experiments in 24 forests across Japan. Environ Health Prev Med. 2010 Jan;15(1):18-26. doi: 10.1007/s12199-009-0086-9. PMID 19568835
- [Background] Park SH, Mattson RH. Ornamental indoor plants in hospital rooms enhanced health outcomes of patients recovering from surgery. J Altern Complement Med. 2009 Sep;15(9):975-80. doi: 10.1089/acm.2009.0075. PMID 19715461
- [Background] Posch M, Bauer P, Brannath W. Issues in designing flexible trials. Stat Med. 2003 Mar 30;22(6):953-69. doi: 10.1002/sim.1455. PMID 12627412
- [Background] Robinson L, Hutchings D, Corner L, Beyer F, Dickinson H, Vanoli A, Finch T, Hughes J, Ballard C, May C, Bond J. A systematic literature review of the effectiveness of non-pharmacological interventions to prevent wandering in dementia and evaluation of the ethical implications and acceptability of their use. Health Technol Assess. 2006 Aug;10(26):iii, ix-108. doi: 10.3310/hta10260. PMID 16849002
- [Background] Ulrich RS. View through a window may influence recovery from surgery. Science. 1984 Apr 27;224(4647):420-1. doi: 10.1126/science.6143402.
- See also: Virtual Reality Aimed At The Elderly Finds New Fans — http://www.npr.org/sections/healthshots/2016/06/29/483790504/virtual-reality-aimed-at-the-elderly-finds-new-fans
- See also: People with dementia test-drive virtual reality rehabilitation system used by injured soldiers to help their condition — http://www.independent.co.uk/life-style/health-and-families/healthnews/dementia-sufferers-test-drive-revolutionary-rehabilitation-system-whichputs-individuals-at-the-helm-of-a6946821.html